CLINICAL TRIAL: NCT03598088
Title: Safety and Acceptability Study of a Non-Hormonal Ring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Daré Bioscience, Inc. (Industry)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: DR-OVP-001; 1R44HD095724-01 (NIH)
Record Dates: First submitted 2018-06-21; First posted 2018-07-26 (Actual); Results first posted 2022-06-08 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Contraception

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Healthy Sexually Active Women (Other): Healthy, sexually active women who are not at risk for pregnancy due to previous female tubal sterilization will receive both Ovaprene and the Caya diaphragm throughout the course of the trial. The purpose of the Caya Post Coital Test (PCT) cycle is to ensure that in this study population and at these sites, results that are expected to be observed in a PCT cycle with an approved vaginal barrier can be replicated.
  Interventions: Device: Ovaprene

INTERVENTIONS:
Device: Ovaprene — non-hormonal contraceptive ring

SUMMARY:
This is a feasibility, multi-center, open-label, non-significant risk device study for a non-hormonal contraceptive ring.

DETAILED DESCRIPTION:
The purpose of this clinical trial is to assess the ability of Ovaprene™ to prevent sperm from penetrating midcycle cervical mucus. In addition, safety, release of ingredients, acceptability and fit will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 18-50 years, inclusive
2. General good health, by volunteer history and per investigator judgment
3. History of regular menstrual cycles of 24-35 days (inclusive), by volunteer report
4. History of Pap tests and follow-up consistent with standard medical practice or willing to undergo a Pap test at Visit 1.
5. Protected from pregnancy by female tubal sterilization
6. Willing to abstain from or engage in intercourse with and without condoms and to abstain from other vaginal activity as required in the protocol
7. In a mutually monogamous relationship for at least the last four months with a male partner who:

   1. Is at least 18 years old;
   2. Has no known risk for Sexually Transmitted Infections (STIs);
   3. Is willing and able to comply with protocol requirements including sexual activity/ abstinence and condom use requirements; and
   4. Can engage in vaginal intercourse with the participant, with and without condoms, as specified in protocol
8. Vaginal and cervical anatomy that, in the opinion of the investigator, lends itself to easy colposcopy and genital tract sample collection
9. Willing to give voluntary consent, sign an informed consent form and comply with study procedures as required by the protocol

Exclusion Criteria:

1. History of hysterectomy
2. Vasectomy in male partner
3. Sterility or known history of sperm dysfunction in male partner
4. Within two calendar months from the last pregnancy outcome. Note: If recently pregnant must have had at least two spontaneous menses since pregnancy outcome.
5. Current use of any hormonal contraceptive or a copper IUD (intra-uterine device), or use of Depo-Provera within the last 120 days
6. Currently breastfeeding or having breastfed an infant in the last two months, or planning to breastfeed during the course of the study
7. Significant gynecological abnormalities (including abnormal vaginal bleeding or excessive vaginal discharge)
8. Either device does not appropriately fit volunteer, as determined by clinician
9. Inability of the volunteer to insert, position, and/or remove either device, even with assistance
10. History of sensitivity/allergy to nonoxynol-9 or to silicone or any other component of Ovaprene™ or Caya, for either the volunteer or her male partner
11. In the last four months, either the volunteer or her male partner diagnosed with or treated for any STI or pelvic inflammatory disease. Note: Women or male partners with a history of genital herpes or condylomata who have been asymptomatic for at least six months may be considered for eligibility
12. Positive test for Trichomonas vaginalis, Neisseria gonorrhea, Chlamydia trachomatis, or HIV
13. Deep epithelial genital findings such as abrasions, ulcerations, and lacerations, or vesicles suspicious for a sexually transmitted infection
14. Chronic or acute vulvar or vaginal symptoms (pain, irritation, spotting, etc.)
15. Known current drug or alcohol abuse which could impact study compliance. (This is defined as any illicit drug use or more than 15 alcoholic drinks per week)
16. Participation in any other investigational trial within the last 30 days or planned participation in any other investigational trial during the study
17. History of gynecological procedures (including genital piercing) on the external genitalia, vagina or cervix within the last 14 days
18. Abnormal finding on laboratory or physical examination or a social or medical condition in either the volunteer or her male partner which, in the opinion of the investigator, would make participation in the study unsafe or would complicate interpretation of data
19. Nugent score greater than or equal to 7
20. Systemic use in the last two weeks or anticipated use during the study of antibiotics (other than those used to treat urinary tract infection (UTI), vaginal candidiasis, or bacterial vaginosis (BV) diagnosed at Visit 1, or to treat UTI or vaginal candidiasis after Visit 1) or topical antivirals (e.g., acyclovir or valacyclovir). Note: Participants should avoid non-steroidal anti-inflammatory drugs (NSAIDs) and Tylenol except for occasional use, as in treatment of headaches or dysmenorrhea.
21. Grade 2 or higher abnormality per the March 2017 update of the Division of AIDS (DAIDS), National Institute of Allergy and Infectious Disease (NIAID) Table for Grading of the Severity of Adverse Events or clinically significant lab abnormalities as determined by the investigator (see Section 13.5 for link to DAIDS table)
22. Inability to achieve adequate cervical mucus in two attempts at the baseline cycle
23. Inadequate sperm in endocervical aspirate during baseline testing without any device, despite adequate mucus and presence of sperm in vaginal pool

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Females and their male partners to be enrolled.
Enrollment: 38 (Actual)
Dates: Start 2018-05-23 (Actual); Primary Completion 2019-10-17 (Actual); Study Completion 2019-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nadene A. Zack, MS, Study Director — Sr Director, Clinical Operations
Locations (6):
- United States (6):
  - University of California at Davis, Sacramento, California
  - Segal Trials, North Miami, Florida
  - Clinical Research Prime, Idaho Falls, Idaho
  - Oregon Health and Science University, Portland, Oregon
  - University of Pennsylvania Penn Obstetric Gynecology Associates, Philadelphia, Pennsylvania
  - Eastern Virginia Medical School, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Sexually Active Women: Healthy, sexually active women who are not at risk for pregnancy due to previous female tubal sterilization will receive both Ovaprene (3 rings over 3 cycles (1 ring per cycle)) and the Caya diaphragm (to be used for intercourse at 1 time for 1 cycle) throughout the course of the trial. Each cycle was 28-35 days long. The purpose of the Caya PCT cycle is to ensure that in this study population and at these sites, results that are expected to be observed in a PCT cycle with an approved vaginal barrier can be replicated.
  Ovaprene: non-hormonal contraceptive ring
Period: Screening/Baseline PCT Visits 1-4
Arm/Group | Healthy Sexually Active Women
Started | 38
Completed | 38
Not Completed | 0
Period: Caya PCT Cycle, Visit 5 & 6
Arm/Group | Healthy Sexually Active Women
Started | 38
Completed | 35
Not Completed | 3
Period: OVP Safety Cycle Visits 7-11
Arm/Group | Healthy Sexually Active Women
Started | 33
Used the OVP Device During the Study | 33 (Any subject that used the OVP device at least one time during the study.)
Completed (2 subjects completed Visit 6, but discontinued prior to Visit 7) | 28
Not Completed | 5
Period: OVP PCT Cycle A Visits 12-16
Arm/Group | Healthy Sexually Active Women
Started | 28
Completed 1 OVP PCT Cycle | 26 (Subjects Completed One PCT Visit)
Completed | 24
Not Completed | 4
Period: OVP PCT Cycle B Visits 17-21
Arm/Group | Healthy Sexually Active Women
Started | 24
Completed | 23
Not Completed | 1

BASELINE CHARACTERISTICS:
Population: All Enrolled Population are those participants that met eligibility criteria.
Groups:
- All Enrolled Population: Healthy, sexually active women who are not at risk for pregnancy due to previous female tubal sterilization will receive both Ovaprene and the Caya diaphragm throughout the course of the trial. The purpose of the Caya PCT cycle is to ensure that in this study population and at these sites, results that are expected to be observed in a PCT cycle with an approved vaginal barrier can be replicated.
Arm/Group | All Enrolled Population
Number analyzed (Participants) | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.8 (6.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 34
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 30
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 38
BMI [Mean (Standard Deviation); unit: kg/m^2] | 29.93 (8.723)

OUTCOME MEASURES:

1. Primary Outcome: Changes From Baseline in the Post Coital Test Results (PCT) Due to Device Use.
Description: All participants had fewer than 5 progressively motile sperm per high power field (PMS/HPF) in all cycles during Ovaprene use.
Time Frame: Baseline to OVP PCTa at 175 Days
Measure: Count of Participants; unit: Participants
Groups:
- Ovaprene Population: All Enrolled Participants that used the Ovaprene device during the study for one PCT cycle.
Arm/Group | Ovaprene Population
Number analyzed (Participants) | 26
Participants
  Number of participants with an Average of Fewer than 5 PMS/HPF in Cervical Mucus at Baseline | 0
  Number of participants with an Average of Fewer than 5 PMS/HPF in Cervical Mucus at OVP3A | 26

2. Other Pre Specified Outcome: Changes in Cervicovaginal pH Pre-coitus and Post-coitus in the Absence of the Study Device.
Description: Evaluating the change in CVF pH before and after sex with no device present.
Time Frame: Pre-Intercourse (Baseline Visit 1) and Post-Intercourse (Baseline Visit 2) (24hrs)
Population: There were 7 subjects that did not have an evaluable result for pH in Cervicovaginal Fluid at these timepoints.
Measure: Mean (Standard Deviation); unit: pH
Groups:
- Ovaprene Population: All Enrolled Participants that used the Ovaprene device during the study.
Arm/Group | Ovaprene Population
Number analyzed (Participants) | 26
pH
  Pre-Intercourse Visit 1 | 6.42 (0.804)
  Post-Intercourse Visit 2 | 6.92 (0.417)

3. Other Pre Specified Outcome: Changes in Cervicovaginal pH Pre-coitus and Post-coitus in the Presence of the Study Device.
Description: Evaluating the change in CVF pH before and after intercourse when the Ovaprene device was being worn during intercourse.
Time Frame: OVP Cycle A Visit 13 (Day 121) to Visit 14 (Day 122) and OVP Cycle B Visit 18 (Day 156) to Visit 19 (Day 157).
Measure: Mean (Standard Deviation); unit: pH
Groups:
- Ovaprene Population, PCT A: All Enrolled Participants that used the Ovaprene device during OVP PCT Cycle A.
- Ovaprene Population, PCT B: All Enrolled Participants that used the Ovaprene device during OVP PCT Cycle B.
Arm/Group | Ovaprene Population, PCT A | Ovaprene Population, PCT B
Number analyzed (Participants) | 26 | 23
pH
  Pre-Intercourse Visit 13 (A) Visit 18 (B) | 6.15 (1.147) | 5.94 (1.266)
  Post-Intercourse Visit 14 (A); Visit 19 (B) | 6.57 (0.890) | 6.40 (1.011)

4. Other Pre Specified Outcome: Incidence of Treatment Emergent Adverse Events (Safety and Tolerability) During Use of the Device.
Description: Number of participants within the Ovaprene population that experienced a Urogenital treatment emergent adverse event (AE).
Time Frame: 175 days
Measure: Count of Participants; unit: Participants
Groups:
- Ovaprene Population: All Enrolled Participants that used the Ovaprene device
Arm/Group | Ovaprene Population
Number analyzed (Participants) | 33
Participants | 21

5. Other Pre Specified Outcome: Number of Participants With Changes in Pelvic Exam Findings From Baseline
Description: Pelvic exams were completed at all 21 visits via a vaginal Colposcopy procedure.
Time Frame: 175 days
Measure: Count of Participants; unit: Participants
Arm/Group | Ovaprene Population
Number analyzed (Participants) | 33
Participants | 0

6. Other Pre Specified Outcome: Changes From Baseline in Nugent Score
Description: Nugent scores were calculated prior to the insertion of each Ovaprene device and then after the device was removed at the end of each cycle.
  Nugent score is a gram stain storage system assessing vaginal bacteria present on a scale of 0-10. Scores ranging from 7-10 are indicative of bacterial vaginosis.
Time Frame: 175 days
Population: Baseline was defined as the first visit of the Ovaprene Cycle (OS1 (Visit 7), OP1a (Visit 12), OP1b (Visit 17)) For Nugent Scores.
  The OS Cycle (Safety cycle) was the 3rd cycle for each participant approximately Days 84 to 105. OPa was the 4th cycle (approximately Days 112 to 140) and OPb was the 5th cycle (approximately days 140 to 175).
Measure: Mean (Standard Deviation); unit: Score (0-10)
Groups:
- Ovaprene Population, Nugent Score: All Enrolled Participants that used the Ovaprene device
Arm/Group | Ovaprene Population, Nugent Score
Number analyzed (Participants) | 33
Score (0-10)
  Change from OS1 to OS2 | 0.8 (1.79)
  Change from OS1 to OS3: number analyzed (Participants) | 31
  Change from OS1 to OS3 | 1.3 (3.16)
  Change from OS1 to OS4: number analyzed (Participants) | 27
  Change from OS1 to OS4 | 1.3 (2.75)
  Change from OS1 to OS5: number analyzed (Participants) | 28
  Change from OS1 to OS5 | 0.9 (2.03)
  Change from OP1A to OP5A: number analyzed (Participants) | 24
  Change from OP1A to OP5A | -0.2 (2.63)
  Change from OP1B to OP5B: number analyzed (Participants) | 24
  Change from OP1B to OP5B | 1.1 (2.59)

7. Other Pre Specified Outcome: Changes From Baseline in Antibacterial (Anti-E. Coli) Activity in Cervicovaginal Fluid.
Description: Measuring the E.coli inhibition (%) pre and post intercourse
Time Frame: Pre Baseline (Day 1) to Post Baseline (Day 2); OVP PCTa Pre Intercourse (Visit 13, Day 121) to Post Intercourse (Visit 14, Day 122) and PCTb Pre Intercourse (Visit 18, Day 156) to Post Intercourse (Visit 19, Day 157).
Population: The number of participants analyzed is based on the number of viable samples collected at each timepoint.
Measure: Mean (Standard Deviation); unit: % inhibition of vaginal bacterial growth
Arm/Group | Ovaprene Population
Number analyzed (Participants) | 33
% inhibition of vaginal bacterial growth
  Baseline Pre-Intercourse (Visit 3): number analyzed (Participants) | 23
  Baseline Pre-Intercourse (Visit 3) | 29.81 (40.16)
  Baseline Post-Intercourse (Visit 4): number analyzed (Participants) | 23
  Baseline Post-Intercourse (Visit 4) | -7.42 (37.54)
  OVPa Pre-Intercourse (Visit 13): number analyzed (Participants) | 27
  OVPa Pre-Intercourse (Visit 13) | 27.23 (47.47)
  OVPa Post-Intercourse (Visit 14): number analyzed (Participants) | 25
  OVPa Post-Intercourse (Visit 14) | 15.66 (46.41)
  OVPb Pre-Intercourse (Visit 18): number analyzed (Participants) | 23
  OVPb Pre-Intercourse (Visit 18) | 28.10 (40.85)
  OVPb Post-Intercourse (Visit 19): number analyzed (Participants) | 23
  OVPb Post-Intercourse (Visit 19) | 10.62 (37.70)

8. Other Pre Specified Outcome: Changes From Baseline in Soluble Markers of Inflammation in Cervicovaginal Fluid.
Description: Measurement of Interleukin-1 Beta (pg IL-1Beta/ug Protein), Interleukin-8 (pg IL-8/ug Protein), Secretory leukocyte Peptidase Inhibitor (SLPI)
Time Frame: as for outcome 7
Population: The number of participants analyzed corresponds to the number of viable samples received for analysis.
Measure: Mean (Standard Deviation); unit: pg/ug
Groups:
- Ovaprene Population, IL-1Beta; Ovaprene Population, IL-8; Ovaprene Population, SLPI: All Enrolled Participants that used the Ovaprene device
Arm/Group | Ovaprene Population, IL-1Beta | Ovaprene Population, IL-8 | Ovaprene Population, SLPI
Number analyzed (Participants) | 33 | 33 | 33
pg/ug
  Baseline Pre-Intercourse (Visit 2): number analyzed (Participants) | 16 | 16 | 16
  Baseline Pre-Intercourse (Visit 2) | 0.075 (0.144) | 2.6563 (7.3156) | 2640.005 (2708.657)
  Baseline Post-Intercourse (Visit 3): number analyzed (Participants) | 16 | 16 | 16
  Baseline Post-Intercourse (Visit 3) | 0.093 (0.192) | 3.3688 (7.9979) | 2175.645 (1895.113)
  OVPa Pre-Intercourse (Visit 13): number analyzed (Participants) | 23 | 23 | 23
  OVPa Pre-Intercourse (Visit 13) | 0.101 (0.134) | 1.2470 (0.8429) | 282.344 (248.081)
  OVPa Post-Intercourse (Visit 14): number analyzed (Participants) | 23 | 23 | 23
  OVPa Post-Intercourse (Visit 14) | 0.111 (0.223) | 0.7870 (0.7914) | 1706.977 (2856.200)
  OVPb Pre-Intercourse (Visit 18): number analyzed (Participants) | 23 | 23 | 23
  OVPb Pre-Intercourse (Visit 18) | 0.119 (0.264) | 1.5135 (1.3988) | 309.313 (411.673)
  OVPb Post-Intercourse (Visit 19): number analyzed (Participants) | 23 | 23 | 22
  OVPb Post-Intercourse (Visit 19) | 0.141 (0.342) | 0.4291 (0.300) | 700.894 (416.64)

9. Other Pre Specified Outcome: Number of Participants With a Study Devices That Has Been Worn for One Cycle With Staphylococcus Aureus Presence on Study Device.
Description: Vaginal samples and swabs of the used Ovaprene devices were tested for growth of staphylococcus aureus.
Time Frame: 35 days (one complete cycle)
Population: Analysis was performed on rings worn for one full cycle.
Measure: Count of Participants; unit: Participants
Arm/Group | Ovaprene Population
Number analyzed (Participants) | 33
Participants | 0

10. Other Pre Specified Outcome: Number of Devices With Presence of Group A Streptococcus That Have Been Worn for One Cycle.
Description: Vaginal samples and swabs of the used Ovaprene devices were tested for group A Streptococcus.
Time Frame: 35 days (one full cyle)
Measure: Count of Participants; unit: Participants
Arm/Group | Ovaprene Population
Number analyzed (Participants) | 33
Participants | 0

11. Other Pre Specified Outcome: Summary of the Acceptability of the Study Device Among Male and Female Participants.
Description: Summary of Open-Ended Acceptability Questionnaire
Time Frame: 175 days
Population: Each participant could answer the questionnaire 3 times, one for each Ovaprene cycle therefore one participant could have made the same comment 3 times. The results display the number of times a comment was made.
  All comments were pooled together in this table.
Measure: Number; unit: participant comments
Units Other Than Participants: Comments Received
Arm/Group | Ovaprene Population
Number analyzed (Participants) | 33
Number analyzed (Comments Received) | 199
participant comments
  Easy to use/insert/convenient | 48
  Not Pericoital | 29
  Does not slip out | 2
  At home removal and insertion | 2
  Comfortable/cannot tell it is there | 52
  Lack of side effects | 9
  Hormone-free | 32
  Discreet, small, light, soft | 17
  Altruism | 4
  Iron supplementation | 1
  Easy for the doctor to take out and put back in | 1
  Learning about how my body changes through different cycles | 1
  I believe its effective | 1

12. Other Pre Specified Outcome: Participants Who Could be Fitted With the Ovaprene Device
Time Frame: Screening or BP3 Visit (2 days)
Measure: Count of Participants; unit: Participants
Groups:
- All Enrolled Population: Healthy, sexually active women who are not at risk for pregnancy due to previous female tubal sterilization.
Arm/Group | All Enrolled Population
Number analyzed (Participants) | 32
Participants | 32

13. Other Pre Specified Outcome: Participants That Could Correctly Insert, Position and Remove the Ovaprene Device
Description: Number of participants that required written instructions, those who required written and verbal instructions and those who needed physical assistance.
Time Frame: Visit 3 (BP3, Day 15-20); Visit 7 (OS1, Day 84); Visit 12 (OP1a, Day 112); Visit 13 (OP2a, Day 122-132); Visit 17 (OP1b, Day 140); UNS could occur at any point during the 175 day study duration
Population: The sites were reminded during a site call on 2/11/2019 that they were to allow patients to try to insert, position, and remove the device using only written instructions. After that point, there were 20 patients who were given the opportunity to do this. Not all participants attempted this at all visits.
Measure: Count of Participants; unit: Participants
Groups:
- Ovaprene Population at BP3; Ovaprene Population at OS1; Ovaprene Population at OP1A; Ovaprene Population at OP2A; Ovaprene Population at OP1B; Ovaprene Population at Unscheduled Visit: All Enrolled Participants that used the Ovaprene device
Arm/Group | Ovaprene Population at BP3 | Ovaprene Population at OS1 | Ovaprene Population at OP1A | Ovaprene Population at OP2A | Ovaprene Population at OP1B | Ovaprene Population at Unscheduled Visit
Number analyzed (Participants) | 15 | 12 | 12 | 1 | 13 | 1
Participants
  Insert - written only | 13 | 12 | 12 | 1 | 13 | 1
  Insert - written and verbal instructions | 2 | 0 | 0 | 0 | 0 | 0
  Insert - physical assistance needed | 0 | 0 | 0 | 0 | 0 | 0
  Position - written only | 12 | 11 | 12 | 1 | 13 | 1
  Position - written and verbal instructions | 3 | 1 | 0 | 0 | 0 | 0
  Position - physical assistance required | 0 | 0 | 0 | 0 | 0 | 0
  Remove - written only: number analyzed (Participants) | 15 | 9 | 8 | 0 | 9 | 1
  Remove - written only | 11 | 9 | 0 | 0 | 9 | 1
  Remove - written and verbal instructions: number analyzed (Participants) | 15 | 9 | 8 | 0 | 9 | 1
  Remove - written and verbal instructions | 4 | 0 | 0 | 0 | 0 | 0
  Remove - physical assistance required: number analyzed (Participants) | 15 | 9 | 8 | 0 | 9 | 1
  Remove - physical assistance required | 0 | 0 | 0 | 0 | 0 | 0

14. Other Pre Specified Outcome: Location of Ovaprene in Relation to Cervix
Description: Location was determined digitally and visually by the investigators.
Time Frame: 175 days
Population: The examinations at Screening were amended to occur at BP3, so later participants only had a check at BP3.
Measure: Count of Participants; unit: Participants
Groups:
- Ovaprene Population at Screening; Ovaprene Population at BP3; Ovaprene Population at OS1; Ovaprene Population at OS2; Ovaprene Population at OS3; Ovaprene Population at OS4; Ovaprene Population at OS5; Ovaprene Population at OP1A; Ovaprene Population at OP2A; Ovaprene Population at OP3A; Ovaprene Population at OP4A; Ovaprene Population at OP5A; Ovaprene Population at OP1B; Ovaprene Population At OP2B; Ovaprene Population at OP3B; Ovaprene Population at OP4B; Ovaprene Population at OP5B: All Enrolled Participants that used the Ovaprene device
Arm/Group | Ovaprene Population at Screening | Ovaprene Population at BP3 | Ovaprene Population at OS1 | Ovaprene Population at OS2 | Ovaprene Population at OS3 | Ovaprene Population at OS4 | Ovaprene Population at OS5 | Ovaprene Population at OP1A | Ovaprene Population at OP2A | Ovaprene Population at OP3A | Ovaprene Population at OP4A | Ovaprene Population at OP5A | Ovaprene Population at OP1B | Ovaprene Population At OP2B | Ovaprene Population at OP3B | Ovaprene Population at OP4B | Ovaprene Population at OP5B
Number analyzed (Participants) | 15 | 17 | 21 | 33 | 32 | 27 | 28 | 26 | 27 | 26 | 26 | 24 | 23 | 24 | 24 | 24 | 24
Participants
  Digital Exam: Over cervical os | 15 | 17 | 21 | 33 | 29 | 26 | 28 | 26 | 25 | 24 | 25 | 23 | 23 | 24 | 24 | 24 | 22
  Digital: not over cervical os - on anterior vaginal wall | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Digital: Not over cervical os/not on anterior vaginal wall | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Visual: Over cervical os | 15 | 17 | 21 | 33 | 30 | 26 | 28 | 26 | 25 | 24 | 25 | 23 | 23 | 24 | 23 | 24 | 22
  Visual: not over cervical os - on anterior vaginal wall | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Visual: Not over cervical os/not on anterior vaginal wall | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 1

ADVERSE EVENTS:
Time Frame: Adverse Event information was collected from time of consent (Screening Visit/Baseline) to Completion (Visit 21); 175 days.
Description: The Caya diaphragm was set up as a control (not a comparator device) to ensure participants could perform a successful Post-Coital Test using a marketed device. The Caya device was only used for 1 act of sexual activity whereas Ovaprene was worn continuously for three 28-day cycles, so the comparison of Adverse Events is not a valid one.
Groups:
- Ovaprene Device: All Enrolled Participants that used the Ovaprene device
- Caya Cycle: All Enrolled Participants that used the Caya diaphragm.
Arm/Group | Ovaprene Device | Caya Cycle
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/35
Other Adverse Events (participants affected / at risk) | 21/33 | 0/35
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ovaprene Device (N=33) | Caya Cycle (N=35)
Bacterial Vaginosis (Infections and infestations) | 8 (9) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 2 (2) | 0 (0)
Adnexa uteri pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Dyspareunia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Merorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pelvic Pain (Reproductive system and breast disorders) | 3 (3) | 0 (0)
Pruritus genital (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Uterine spasm (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Vaginal Discharge (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Post procedural hemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0) — spotting due to having to use tenaculum to see cervix
Vaginal Odor (Reproductive system and breast disorders) | 9 (11) | 0 (0)
Vulvar Erosion (Reproductive system and breast disorders) | 1 (2) | 0 (0)
Vulvovaginal dryness (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 2 (2) | 0 (0)
dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Hemorrhage (Vascular disorders) | 1 (1) | 0 (0) — Intermittent bleeding (non-menses)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PIs are restricted from publishing results without prior approval from the Sponsor.

DOCUMENTS (2):
  • Study Protocol (2019-06-13): https://cdn.clinicaltrials.gov/large-docs/88/NCT03598088/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-06): https://cdn.clinicaltrials.gov/large-docs/88/NCT03598088/SAP_001.pdf